CLINICAL TRIAL: NCT06500000
Title: The Plasma Metabolomics Profiling of Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Other Study IDs: MP of PA
Record Dates: First submitted 2024-06-30; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Primary Aldosteronism; Essential Hypertension; Idiopathic Aldosteronism; Aldosterone-producing Adenoma
MeSH Terms: conditions — Hyperaldosteronism; Essential Hypertension; Adrenocortical Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- essential hypertension (EH): According to 2010 Chinese guidelines for the management of essential hypertension (EH), EH was defined as systolic BP (SBP) ≥140 mm Hg, diastolic BP (DBP) ≥90 mm Hg, and use of antihypertensive medicine within 2 weeks and excluded from PA through ARR or diagnostic testing.
  Interventions: Diagnostic Test: liquid chromatography-mass spectrometry (LC/MS)
- idiopathic aldosteronism (IHA): Patients were confirmed to be diagnosed with primary aldosteronism (PA) in accordance with the Endocrine Society Clinical Practice Guideline criteria. Antihypertensive drugs that may affect the renin-angiotensin-aldosterone system (RAAS) were discontinued for at least 2-4 weeks. Patients with an aldosterone-to-renin ratio (ARR) > 3.7 (ng/dL) further underwent one of the following confirmatory tests: saline infusion test (infusion of 2 L isotonic saline within 4 h) or captopril-inhibition test (oral administration of 50 mg captopril). Adrenal CT scan and adrenal vein sampling (AVS) were performed for PA subtype classification. Patients with IHA were determined based on the absence of obvious adenoma on adrenal CT and bilateral aldosterone overproduction.
  Interventions: Diagnostic Test: liquid chromatography-mass spectrometry (LC/MS)
- aldosterone-producing adenoma (APA): Patients were confirmed to be diagnosed with primary aldosteronism (PA) in accordance with the Endocrine Society Clinical Practice Guideline criteria. Antihypertensive drugs that may affect the renin-angiotensin-aldosterone system (RAAS) were discontinued for at least 2-4 weeks. Patients with an aldosterone-to-renin ratio (ARR) > 3.7 (ng/dL) further underwent one of the following confirmatory tests: saline infusion test (infusion of 2 L isotonic saline within 4 h) or captopril-inhibition test (oral administration of 50 mg captopril). Adrenal CT scan and adrenal vein sampling (AVS) were performed for PA subtype classification. Patients with APA were identified based on macroadenoma >1 cm on adrenal CT, unilateral hypersecretion of aldosterone, and pathological confirmation.
  Interventions: Diagnostic Test: liquid chromatography-mass spectrometry (LC/MS)

INTERVENTIONS:
Diagnostic Test: liquid chromatography-mass spectrometry (LC/MS) — Metabolomics is a rapidly evolving high-throughput technology that allows the measurement of the entire complement of metabolites generated by biochemical reactions under certain conditions in biological fluids or tissues. This technology has been used extensively to identify biomarkers in various cancers, nervous system diseases, cardiovascular diseases, pituitary diseases, and other diseases. The identification of biomarkers can be clinically useful for a more accurate diagnosis, prognosis, and treatment choice as well as disease monitoring. Among mass spectrometry (MS) methods, liquid chromatography- mass spectrometry (LC-MS) has been recognized as a robust metabolomics tool and has been widely applied in metabolite identification and quantification due to its high sensitivity, peak resolution, and reproducibility.

SUMMARY:
Primary aldosteronism (PA), characterized by overt renin-independent aldosterone production, is the most common form endocrine hypertension. Compared with blood pressure-matched cases of essential hypertension (EH), PA is associated with a higher risk of cardiovascular morbidity and mortality. It is estimated that PA affects at least 10% of hypertensive patients and up to 25% of treatment-resistant hypertension. The major subtypes of PA are comprised of bilateral idiopathic hyperaldosteronism (IHA) and unilateral aldosterone-producing adenoma (APA). The screening, confirmatory testing, and subtype differentiation of PA for therapeutic management is a multi-step and complex process, resulting in low screening rates and poor clinical recognition.

PA is an independent risk factor for metabolic morbidity. Metabolomic profiling is a relatively new strategy for the diagnosis and prognosis of disease through identification and quantification of various metabolites. In the current study, we aimed to investigate the potential biomakers for discriminating PA from EH, as well as subtype classification for PA, by untargeted metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* According to 2010 Chinese guidelines for the management of Essential hypertension (EH), EH was defined as systolic blood pressure (SBP) ≥140 mm Hg, diastolic blood pressure (DBP) ≥90 mm Hg, and use of antihypertensive medicine within 2 weeks and excluded from PA through ARR or confirmatory testing.
* Patients were confirmed to be diagnosed with Primary aldosteronism (PA) in accordance with the Endocrine Society Clinical Practice Guideline criteria. Patients with an aldosterone-to-renin ratio (ARR) > 3.7 (ng/dL) further conformed with one of the following confirmatory tests: saline infusion test or captopril-inhibition test. Adrenal CT scans and Adrenal venous sampling (AVS) were performed for PA subtype classification.
* Patients with idiopathic hyperaldosteronism (IHA) were determined based on the absence of obvious adenoma on adrenal CT and bilateral aldosterone overproduction.
* Patients with aldosterone-producing adenoma (APA) were identified based on macroadenoma >1 cm on adrenal CT, unilateral hypersecretion of aldosterone, and pathological confirmation.
* Signed informed consent and agreed to participate in this study.

Exclusion Criteria:

* other subtypes of secondary hypertension, including renal hypertension, renovascular hypertension, and adrenal hypertension (i.e., pheochromocytoma and Cushing syndrome).
* adrenal cortical carcinoma
* acute infection at the time of assessment
* severe cardiovascular or cerebrovascular disease, liver or renal dysfunction, tumors, autoimmune disease or mental disorders.
* history of adrenalectomy
* alcohol abuse or pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 75 hypertensive patients diagnosed with PA and 20 additional age-, sex-, body mass index (BMI)- and waist circumference- matched essential hypertensive patients were recruited from the Department of Hypertension and Endocrinology, Army Medical Center, Army Medical University, Chongqing, China, from August to October 2022. Informed consent was obtained from each participant.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
The potential biomarkers for primary aldosteronism diagnosis via untargeted metabolomics | 4 months
  The differentially expressed metabolites between primary aldosteronism (PA) and essential hypertension (EH) will be identified by untargeted metabolomics. The differentially expressed metabolites with good discriminative capability for determination of PA from EH can serve as biomarkers for PA diagnosis.
The potential biomarkers for primary aldosteronism subtype classification via untargeted metabolomics | 4 months
  The differentially expressed metabolites between idiopathic aldosteronism (IHA) and aldosterone-producing adenoma (APA) will be identified by untargeted metabolomics. The differentially expressed metabolites with good discriminative capability for determination of APA from IHA can serve as biomarkers for PA subtype classification.
The predictive models for PA diagnosis and subtype classification by machine learning | 4 months
  The predictive models will be constructed through the application of machine learning, integrating clinical data with differentially expressed metabolites for the diagnosis and subtype classification of PA

CONTACTS AND LOCATIONS:
Locations (1):
- China Chongqing The third hospital affiliated to the Third Millitary Medical University, Chongqing, Chongqing Municipality, China